CLINICAL TRIAL: NCT01861964
Title: Effects of Xylooligosarcharide on Composition of the Human Colonic Microflora
Acronym: XOS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: LBIXOS001
Record Dates: First submitted 2013-05-08; First posted 2013-05-24 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Bifidobacteria; Healthy Volunteers
Keywords: XOS; Xylooligosarcharide; Prebiotic
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sugar Pill (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo (Maltodextrin)
- Xylooligosarcharide 2.8g (Active Comparator): Xylooligosarcharide 2.8grams
  Interventions: Dietary Supplement: Xylooligosarcharide 2.8g
- Xylooligosarcharide 1.4g (Active Comparator)
  Interventions: Dietary Supplement: Xylooligosarcharide 1.4g

INTERVENTIONS:
Dietary Supplement: Placebo (Maltodextrin) — Maltodextrin 505mg/capsule 8 capsules/day (4 with breakfast and 4 with dinner meal)
  Other Names: Maltodextrin
  Arms: Sugar Pill
Dietary Supplement: Xylooligosarcharide 1.4g — 8 capsules (512 mg/capsule) 4 with breakfast and 4 with dinner meal
  Other Names: XOS 1.4g
  Arms: Xylooligosarcharide 1.4g
Dietary Supplement: Xylooligosarcharide 2.8g — 8 capsules (520 mg/capsule) to be taken in the morning and in the evening
  Other Names: XOS 2.8g
  Arms: Xylooligosarcharide 2.8g

SUMMARY:
Human and animal studies demonstrate that xylooligosaccharides (XOS) are a highly efficacious prebiotic ingredient that delivers benefits at a minimum level of 1.4 g/day (d), which is much lower than levels required by fructooligosaccharides (FOS, 5 g/d) or galactooligosaccharides (GOS, 8 g/d). XOS promotes gastrointestinal regularity and relieves diarrhea and constipation at 0.7 g/d and 1.4 g/d, respectively. Xylooligosaccharides may also reduce blood cholesterol and may improve glycemic control, although more data from clinical trials are needed to confirm preliminary findings.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-50 years of age at screen.
2. In generally good health
3. Subjects must read and sign the Institutional Review Board-approved written informed consent prior to the initiation of any study specific procedures or enrollment. A subject will be excluded for any condition that might compromise the ability to give truly informed consent.

Exclusion Criteria:

1. Any history of gastrointestinal disease except for appendectomy
2. No antibiotic, pre- or probiotic or laxative use during the 2 months before the study.
3. Any subject with a history of diabetes mellitus, or other serious medical condition, such as chronic hepatic or renal disease, bleeding disorder, congestive heart disease, chronic diarrhea disorders, myocardial infarction, coronary artery bypass graft, angioplasty within 6 months prior to screening, current diagnosis of uncontrolled hypertension (defined as systolic BP>160mmHg, diastolic BP>95mmHg), active or chronic gastrointestinal disorders, bulimia, anorexia, or endocrine diseases (except thyroid disease requiring medication) as indicated by medical history or routine physical examination.
4. Any subject with a screening laboratory value outside of the laboratory normal range that is considered clinically significant for study participation by the investigator.
5. Any subject who currently uses tobacco products.
6. Any subject who is pregnant or lactating, or becomes pregnant during the study.
7. Any subject who is unable or unwilling to comply with the study protocol.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The Effects of Xyloologosarcharide (XOS) on colonic bifidobacteria counts in healthy volunteers. | 10 weeks
  After a 2 weeks of run-in, 30 healthy volunteers were randomly assigned to take 1.4 grams/day of XOS, or 2.8 grams/day or placebo for 8 weeks. The bifidobarteria counts was assessed at screening, baseline, 4, 8 weeks on supplementation of XOS and after 2 week cessation of XOS.

SECONDARY OUTCOMES:
Tolerance of XOS by healthy volunteers | 10 weeks
  The tolerance of XOS was assessed by questionnaires, adverse event logs with comparison with placebo control group

CONTACTS AND LOCATIONS:
Overall Officials: David Heber, MD, PhD, Principal Investigator — UCLA Center for Human Nutrition
Locations (2):
- United States (2):
  - UCLA Center for Human Nutriiton, Los Angeles, California
  - UCLA Center for Human Nutrition, David Geffen School of Medicine, Los Angeles, California

REFERENCES:
- [Result] Finegold SM, Li Z, Summanen PH, Downes J, Thames G, Corbett K, Dowd S, Krak M, Heber D. Xylooligosaccharide increases bifidobacteria but not lactobacilli in human gut microbiota. Food Funct. 2014 Mar;5(3):436-45. doi: 10.1039/c3fo60348b. PMID 24513849